CLINICAL TRIAL: NCT03407586
Title: Changing the STI Care Model to Reduce Genital Inflammation and HIV Risk in South African Women
Brief Title: STI Care Model to Reduce Genital Inflammation and HIV Risk in South African Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for the AIDS Programme of Research in South Africa (Network)
Collaborators: Johns Hopkins University (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Dr Nigel Garrett, Head of Pathogenesis and Vaccine Research, Centre for the AIDS Programme of Research in South Africa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CAPRISA 083; R21AI116759 (NIH)
Record Dates: First submitted 2018-01-09; First posted 2018-01-23 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: HIV Prevention; Sexually Transmitted Diseases
Keywords: point-of-care testing; sexually transmitted infections; expedited partner therapy; genital inflammation
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Masking Description: All participants provided written informed consent to join the intervention of diagnostic rather than syndromic management.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic STI care (Other): All participants underwent point-of-care STI testing, and if diagnosed with a STI were offered immediate therapy, and expedited therapy if indicated.
  Interventions: Diagnostic Test: Point-of-care STI testing

INTERVENTIONS:
Diagnostic Test: Point-of-care STI testing — All participants underwent point-of-care STI testing (GeneXpert), and if diagnosed with a STI were offered immediate therapy, and expedited therapy, if indicated.

SUMMARY:
The goal of this prospective cohort study is to determine if a model of care including point-of-care testing, immediate therapy, expedited partner therapy and test of cure will result in a higher cure rate and a lower recurrence rate of sexually transmitted infections (STIs), with a subsequent reduction in genital inflammatory cytokines and hence HIV risk among young women in a high burden setting in KwaZulu-Natal, South Africa. The study will identify individuals with STIs using the GeneXpert system for the simultaneous detection of Neisseria gonorrhoeae and Chlamydia trachomatis, and Trichomonas vaginalis. Genital tract cytokines will be measured using Bio-Plex Pro Human Cytokine kits and a Bio-Plex MagPix Array Reader. Following point-of-care diagnosis, participants will be treated immediately with appropriate therapy under direct supervision, offering the participants expedited partner therapy for their partners. STI testing and cytokine assessments will be repeated after 6 and 12 weeks, to determine if these have decreased. Overall, this study will provide some evidence on whether this STI care model can have an impact on STI prevalence and genital tract inflammation, in a low- and middle-income country, where currently syndromic STI management is the standard of care.

DETAILED DESCRIPTION:
Sexually transmitted infections (STIs) are strongly associated with HIV risk. However, population based studies to manage STIs as a way of reducing HIV risk have had limited success. Recent studies show that elevated genital tract inflammatory cytokines are strongly associated with an increased risk of HIV acquisition, and STIs are one of the commonest causes of elevated genital tract cytokines. This interest in the role of cytokines in HIV acquisition has reinvigorated interest in STIs and whether better management strategies can have a role to play in HIV risk reduction.

HIV and STIs are extremely common in the South African province of KwaZulu-Natal, where there are many challenges with STI diagnosis and treatment, including the reliance on syndromic management, an approach based on the recognition of STI syndromes (vaginal discharge, urethral discharge and genital ulceration), followed by treatment targeting the common causes of the syndrome. This syndromic management approach has a low sensitivity and specificity for detecting the most common curable STIs, such as chlamydia, gonorrhoea, trichomoniasis and syphilis. Studies have shown that only 13% of symptomatic STI infections are cured with the STI treatment services currently offered in KwaZulu-Natal. This low cure rate for symptomatic STIs is compounded by the fact that up to 80% of STIs are asymptomatic, which results in a majority of STIs remaining undiagnosed and untreated. Other challenges with current STI management include limited partner notification and treatment, resulting in high levels of reinfection. At a population level, the result is that most STIs remain untreated and the burden of STIs within the community remains unchecked.

The goal of the study is to determine if an innovative, enhanced programme of STI management will result in a higher cure rate and a lower recurrence rate, with a subsequent reduction in genital inflammatory cytokines and hence HIV risk. This proof-of-concept cohort study will identify individuals with STIs using an innovative, point-of-care diagnostic test, an automated, cartridge-based nucleic amplification assay (GeneXpert) for the simultaneous detection of Neisseria gonorrhoeae and Chlamydia trachomatis, and Trichomonas vaginalis. This technology has been introduced on a large scale across South Africa to detect tuberculosis (TB) and TB drug resistance, thereby accelerating diagnosis, treatment and enhancing public health initiatives to control TB. Genital tract cytokines will be measured using Bio-Plex Pro Human Cytokine kits and a Bio-Plex MagPix Array Reader. Following point-of-care diagnosis, participants will be treated immediately with appropriate therapy under direct supervision, giving the participants the same treatment to take home for their sexual partners (expedited partner therapy) and asking them to return after six weeks and three months for a test of cure and additional cytokine assessments, to determine if these have decreased.

Overall, this innovative enhanced management package for targeted STI care, offers the best opportunity to reduce STIs, by ensuring that the individual is cured and by reducing the risk of reinfection using expedited partner therapy. This will allow the investigators to determine whether genital inflammation can be reduced after effective targeted STI treatment, and ultimately reduce the risk of HIV acquisition in South Africa.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 40 years
* Female gender
* HIV negative antibody test at enrollment

Exclusion Criteria:

* HIV positive women
* Pregnant women
* Women who have had antibiotic treatment within the last 7 days
* Women who disclose any form of sex work

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 267 (Actual)
Dates: Start 2016-05-15 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Changes in genital inflammation in women diagnosed with STIs after a diagnostic care intervention | Baseline and 6 and 12 weeks after the intervention
  Genital cytokine measurements before and after the intervention

SECONDARY OUTCOMES:
Prevalence of laboratory-diagnosed STIs in women presenting to the Prince Cyril Zulu Communicable Diseases Clinic, Durban, South Africa | Baseline
  Prevalence of chlamydia, gonorrhoea and trichomoniasis in young women presenting for syndromic STI care
Validation of GeneXpert technology for STI testing against laboratory-based STI assays | Baseline
  GeneXpert validation
Acceptability of implementing expedited partner therapy among patients | 6 weeks and 3 months after intervention
  Proportion of patients taking up expedited partner therapy

CONTACTS AND LOCATIONS:
Overall Officials: Nigel J Garrett, MBBS, Principal Investigator — Centre for the AIDS Programme of Research in South Africa; Anne Rompalo, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- CAPRISA, Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Data will be published in open access journal together with manuscript, and will thereby be shared with other researchers.
Supporting Information: Study Protocol, SAP
Time Frame: The manuscript and supporting information are currently under review at PLOS ONE journal and are expected to be published indefinitely by 31 January 2018.

REFERENCES:
- [Derived] Garrett N, Mitchev N, Osman F, Naidoo J, Dorward J, Singh R, Ngobese H, Rompalo A, Mlisana K, Mindel A. Diagnostic accuracy of the Xpert CT/NG and OSOM Trichomonas Rapid assays for point-of-care STI testing among young women in South Africa: a cross-sectional study. BMJ Open. 2019 Feb 19;9(2):e026888. doi: 10.1136/bmjopen-2018-026888. PMID 30782948